Originally developed: 1/12 2020

Does Manual Treatment With Craniosacral Therapy Change the Experience of Dry Mouth in People Who Suffers From Dry Mouth After Cancer in Throat Or Mouth - a Pilot Study

NCT05882890

Participants in the research project have been using a standard informed consent form in Danish made by Danish Research Ethics Committees:

Participation in a Health science Research project

Titel of research project: Efficacy of Manual treatment of Tissue in the Diaphragm, Throat, Neck, Cranium and Mouth Region for Radiation-induced Xerostomia and Hypo- or Subnormal Salivation - a case study

(title is later changed to: Does Manuel Treatment With Craniosacral Therapy Change the Experience of Dry Mouth in People Who Suffers With Dry Mouth After Cancer in Throat Ore Mouth - a Pilot Study

Declaration from the participant:

I have received oral and written information and I know enough about purpose, method, benefits and disadvantages to give my yes to participate in this project.

I know that it is <u>voluntarily to participate</u> and that I can always pull back my consent, without loosing my rights for treament now and in the future.

I give my consent to participate in this research project /trial and have received a copy of this consent form and a copy of the written information about the project for private use.

Name of the participant: -----

| Date Signature |
|---|
| Do you want to receive information about the results of the project and any consequences it could have for you |
| yes no |
| Declaration from the person that gives information about the project: |
| I declare, that the participant has received oral and written information about the trial |
| To the best of my knowledge there has been given adequate information, so that the participant can make a decision about participation in this trial |
| Name of the person who gave the information: Cathrine Rahbek |
| Date Signature |